CLINICAL TRIAL: NCT02715102
Title: Determination of the Utility of Plasma Circulating Tumor DNA (ctDNA) Measurements for Detection of Lung Cancer in Patients Undergoing Diagnostic or Therapeutic Bronchoscopy or Thoracotomy
Brief Title: Circulating Tumor DNA in Patients at High Risk for Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Patient accrual was slow due to exclusion of patients with prior cancers
Sponsor: Pathway Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: Pathway Genomics - 006
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Cancer of the Lung; Lung Cancer; Lung Neoplasms; Adenocarcinoma of the Lung; Non Small Cell Carcinoma of the Lung; Small Cell Carcinoma of the Lung
Keywords: lung cancer; lung neoplasms; lung nodules; screening tests for cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted and run in the ctDNA assay. Patients will be asked to either consent or not to consent to having their DNA extracted from the original specimen and their clinical information kept for optional anonymized medical research in the future.
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who are about to undergo a diagnostic or therapeutic bronchoscopy or thoracic surgery without a distant history of cancer will have their blood drawn for measurement of circulating tumor DNA (ctDNA) to validate the utility of molecular diagnostic assays for the early detection of lung cancer.

DETAILED DESCRIPTION:
Specific somatic (i.e. acquired and not inherited) mutations have been found in many cancers. Some of these cancers shed this DNA into the patient's blood stream and is called circulating tumor DNA (ctDNA). Pathway Genomics has developed a new molecular assay that uses blood plasma as the source of DNA fragments. The ctDNA is isolated, amplified and analyzed for the presence of one or more of 96 known mutations that are found in 9 cancer driver genes. This technique of using a "liquid biopsy" to screen for and monitor cancer has been documented in a number of recent medical publications. However, the majority of published studies are on subjects who have already been diagnosed with cancer. Therefore, the investigators wish to look at a population of patients who are scheduled to undergo a diagnostic or therapeutic bronchoscopy or thoracotomy without a know history of cancer (other than basal cell carcinomas of the skin). The blood will be drawn at the time of or a few weeks before the procedure. The analysis of the blood sample will take placed in the Pathway Genomics clinical laboratory which is Clinical Laboratory Improvement Amendments of 1988 (CLIA) certified.

Following an informed consent process, the patients will fill out a health questionnaire and will have the blood drawn prior to the surgical procedure. Up to 30 ml of blood (approximately 2 tablespoons) will be drawn at any one time. The patient will be asked to agree to being contacted by the investigators yearly for up to 5 years to provide follow-up medical information. No patient will be identified in presentations or publications resulting from this work and all data will be reported from analysis of combined information from participants in this study.

Individuals may participate in this study if they are 18 years of age or older, have not had a prior diagnosis of cancer (other than a skin cancer or if they are undergoing the thoracic surgical procedure for a cancer that was diagnosed within the prior month), and are undergoing a diagnostic or therapeutic bronchoscopy or thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, not previously diagnosed with cancer (except for basal cell carcinomas of the skin or a diagnosis of cancer within a month of surgery and for which the surgical procedure is being performed).

Exclusion Criteria:

* Prior history of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to undergo a diagnostic or therapeutic bronchoscopy or thoracotomy by Dr. Robert McKenna.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with lung cancer who had a positive ctDNA result (true positive) | 5 years
  ctDNA results will be correlated with pathology and subsequent clinical findings.

SECONDARY OUTCOMES:
Percentage of patients who develop any cancer during the 5 years of follow-up | 5 years
  ctDNA results will be correlated with pathology and subsequent clinical findings.
Percentage of patients without lung cancer who had a positive ctDNA result (false positive) | 5 years
  ctDNA results will be correlated with pathology and subsequent clinical findings.
Percentage of patients with lung cancer who had a negative ctDNA result (false negative) | 5 years
  ctDNA results will be correlated with pathology and subsequent clinical findings.
Percentage of patients without lung cancer who had a negative ctDNA result (true negative) | 5 years
  ctDNA results will be correlated with pathology and subsequent clinical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. McKenna, M.D., Principal Investigator — Providence Saint John's Health Center
Locations (1):
- Cardiothoracic Outpatient Clinic, Providence Saint John's Health Center, 2121 Santa Monica Blvd., Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Through presentations at scientific meetings and in the peer-reviewed medical literature.